CLINICAL TRIAL: NCT07273526
Title: Comparison of the Efficacy of Renaline and Dopamine in the Treatment of Fluid Refractory Septic Shock in Children
Brief Title: Adrenaline V/s Dopamine in Fuid Refractory Septic Shock
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laiba Qamar (Other)
Responsible Party: Sponsor-Investigator, Laiba Qamar, Sponsor Investigator, University of Health Sciences Lahore
Organization: University of Health Sciences Lahore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #AVDSSC24#
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Fluid Refractory Septic Shock; Septic Shock
Keywords: Septic Shock; Adrenaine; Dopamine; Fluid refractory septic shock
MeSH Terms: conditions — Shock, Septic | interventions — Epinephrine; Dopamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): These patients will receive 0.1-0.3ug/kg/min of adrenaline when diagnosed with fluid refractory Septic shock .
  Interventions: Drug: Adrenaline
- Group B (Active Comparator): The patients in this arm of study will be provided with dopamine 10-20ug/kg/min when diagnosed with fluid refractory septic shock.
  Interventions: Drug: Dopamine

INTERVENTIONS:
Drug: Adrenaline — The adrenaline will be given as a vasoconstrictor in the dose of 0.1-0.3ug/kg/min to the patients in group A when diagnosed with fluid refractory septic shock
  Arms: Group A
Drug: Dopamine — The drug dopamine will be adminitered in dose of 10-20ug/kg/min to the patients of group B when diagnosed with fluid refractory septic shock.
  Arms: Group B

SUMMARY:
This study compares the efficacy of two drugs i.e Adrenaline and dopamine in fluid refractory type of septic shock which is a dreadful medical condition especially in children. The efficacy will be checked based on heart rate , GCS, capillary refill time , palpable pripheral pulse , urine output and systolic blood pressure.

DETAILED DESCRIPTION:
This is a randomized control trial in which children / patients diagnosed with Fluid refractory Septic shock will be provided with one of the two drugs ina randomzied way and their efficacy will be assesed on the basis of correction of various parameters at various points of time.

ELIGIBILITY:
Inclusion Criteria:

Patients of both Genders having age range between 1month and 12 years with diagnosis of fluid refractory septic shock as per operational definition.

-

Exclusion Criteria:

* Patients with

  1. cardiopumonary Bypass during last 5 days
  2. Chronic Systemic disease like Chronic kidney Disease , cerebral palsy, congenital heart disease
  3. neuromuscular discorder
  4. Metabolic disorders
  5. Those who already had treatment at periphery for hypovolemia without any record of medication or sequential organ failure at presentation

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | 6 hours
  The blood pressure of the patients will be meaures after administration of each drug at 20 mins and 6 hours.
Pulse | 6 hours
  The pulse will be compared after adminitration of both drugs at 20 mins and 6 hours
Capillary Refill Time | 6 Hours
  Capillary Refill time will be assessed after administration of each drug at 20 mins and 6 hours
Urine output | 6 hours
  Urine output will be calculated from the time of administration of each drug at 20mins and 6 hours and comapred.
GCS | 6 hours
  Glascow Comma Scale (GCS) will be asses at 20 mins and 6 hours after administration of each drug

SECONDARY OUTCOMES:
SOFA ( Sequential Organ Failure Assesment) | 6 Hours
  SOFA ( Sequential Organ Failure Assesment) score will be calculated afte adminitration of each drug at 20mins and 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- The Children Hospital and The Institute of Child Health Faisalabad, Faisalābad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No